CLINICAL TRIAL: NCT01899053
Title: A Multicenter, Open-label, Phase 1b Study of MLN0128 (an Oral mTORC1/2 Inhibitor) in Combination With MLN1117 (an Oral PI3Kα Inhibitor) in Adult Patients With Advanced Nonhematologic Malignancies
Brief Title: A Safety and Pharmacokinetic Study of TAK-228 in Combination With TAK-117 in Adult Participants With Advanced Nonhematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C32001; 2013-000466-11 (EudraCT Number)
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Advanced Nonhematologic Malignancies
Keywords: Drug Therapy; TAK-228; TAK-117
MeSH Terms: interventions — sapanisertib; serabelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Treatment Arm A (Experimental): TAK-228 2 or 4 mg, capsule (milled or unmilled), orally, once daily every day (QD), and TAK-117 100, 200 or 300 mg, capsule, orally, once on Monday, Wednesday and Friday each week (MWF QW) for up to 13 cycles (each cycle was 28 days), up to approximately 52 weeks.
  Interventions: Drug: TAK-228; Drug: TAK-117
- Dose Escalation Treatment Arm B (Experimental): TAK-228 3, 4, 6 or 8 mg, capsule (milled or unmilled), orally, once on Monday, Tuesday and Wednesday each week (MTuW QW), and TAK-117 100 or 200 mg, capsule, orally, once on MTuW QW for up to 9 cycles (each cycle was 28 days), up to approximately 38.7 weeks.
  Interventions: Drug: TAK-228; Drug: TAK-117
- Dose Escalation Treatment Arm C (Experimental): TAK-228 3 mg, capsule (milled or unmilled), orally, once on MTuW QW, and TAK-117 300 or 400 mg, capsule, orally, once on MTuW QW for up to 17 cycles (each cycle was 28 days), up to approximately 64.3 weeks.
  Interventions: Drug: TAK-228; Drug: TAK-117
- Drug-Drug Interaction (DDI) Expansion Cohort (Experimental): TAK-228 4 mg, capsule (milled), orally, once on MTuW QW except on Days 15, 16 and 17 of Cycle 1, and TAK-117 200 mg, capsule, orally, once on MTuW QW except on Days 1, 2 and 3 of Cycle 1 for up to 8 cycles (each cycle was 28 days), up to approximately 31.4 weeks.
  Interventions: Drug: TAK-228; Drug: TAK-117

INTERVENTIONS:
Drug: TAK-228 — TAK-228 Capsules
  Other Names: MLN0128, INK128 or Sapanisertib
Drug: TAK-117 — TAK-117 Capsules
  Other Names: MLN1117

SUMMARY:
The purpose of this study was to evaluate the safety and to determine dose-limiting toxicities (DLTs), maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D), and dosing schedules of oral TAK-228+TAK-117. It also evaluated the single- and multiple-dose plasma pharmacokinetics (PK) of TAK-228+TAK-117 in participants with advanced nonhematologic malignancies.

DETAILED DESCRIPTION:
The drug being tested in this study was TAK-228. TAK-228 was tested to evaluate the safety, pharmacokinetics and efficacy, of TAK-228 in combination with TAK-117 when administered to adult participants with advanced nonhematologic malignancies.

The study enrolled 101 patients. The study consisted of 2 phases: an escalation stage followed by an expansion stage. Participants in escalation stage were assigned to the following treatment arms:

* Dose escalation treatment arm A: TAK-228 2 or 4 mg capsule
* Dose escalation treatment arm B: TAK-228 3, 4, 6 or 8 mg capsule
* Dose escalation treatment arm C: TAK-228 3 mg capsule

Upon completion of the escalation stage, 1 combination treatment regimen was selected for further safety, tolerability, pharmacokinetics, and mutual drug-drug interaction characterization in the expansion stage. During treatment, participants in both stages received TAK-228 and TAK-117 capsules at prespecified doses in repeated 28-day cycles.

This multi-center trial conducted in the United States, United Kingdom and Spain. The overall time to participate in this study was approximately 68 weeks. Participants made multiple visits to the clinic, and a final visit after 30 days after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years or older
* Participants must have a diagnosis and documented disease progression of a solid tumor malignancy, excluding primary brain tumor, for which standard, curative, or life prolonging treatment does not exist or is no longer effective
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Female participants who are postmenopausal for at least 1 year prior to screening. For women of child-bearing potential agree to practice 2 effective methods of contraception or agree to practice true abstinence
* Male participants must agree to practice effective barrier contraception during the entire study treatment period and through 30 days after last dose of study drug or practice true abstinence
* Voluntary written consent
* Suitable venous access
* Participants must have a block of banked tumor tissue and/or fresh tumor tissue or at least 10 unstained slides available to be sent to the central laboratory
* Clinical laboratory values as specified in the protocol
* Participants must have radiographically or clinically evaluable tumor

Exclusion Criteria:

* Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 before first dose of study drug
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment
* Treatment with any investigational products within 30 days before the first dose of study drug
* Previous treatment with TAK-117 and/or TAK-228; previous treatment with dual mTORC1/2 or dual PI3K-mTOR inhibitors
* Failed to have recovered from the reversible effects of previous anticancer therapies
* Have received systemic corticosteroid (inhalers are allowed) within 7 days before the first administration of study drug
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of study drug
* Diagnosis of diabetes mellitus
* Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active CNS disease, active infection
* Known human immunodeficiency virus (HIV) infection
* Cardiovascular conditions as defined in the protocol
* A requirement for positive inotropic support (excluding digoxin) or serious uncontrolled cardiac arrhythmia (including atrial flutter/fibrillation) within 1 year before screening
* Participants who are taking proton pump inhibitors within 7 days of the first dose or who require treatment with proton pump inhibitors during the trial or those who are taking histamine-2 (H2) receptor antagonists within 24 hours of the first dose
* Participants who received previous therapy with PI3K inhibitors or rapalogs will be allowed in the study if all other inclusion/exclusion criteria are met
* Diagnosis of primary brain tumor or symptomatic brain metastasis. Participants with brain metastases must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events (AEs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-06-28 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (5):
- United States (3):
  - Boston, Massachusetts
  - Nashville, Tennessee
  - San Antonio, Texas
- Barcelona, Spain
- Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in Spain, United Kingdom and United States from 28 June 2013 to 30 April 2018.
Pre-assignment Details: Participants with a diagnosis of advanced nonhematologic malignancies were enrolled. A total of 101 participants were enrolled, out of which 81 entered the escalation phase, and 20 entered the expansion phase.
Groups:
- Dose Escalation Treatment Arm A: Cohort 1A: TAK-228 2 mg, capsule (unmilled), orally, once daily every day (QD), and TAK-117 100 mg, capsule, orally, once on Monday, Wednesday and Friday each week (MWF QW) for up to 4 cycles (each cycle was 28 days), up to 16 weeks.
- Dose Escalation Treatment Arm A: Cohort 2A: TAK-228 4 mg, capsule (unmilled), orally, once daily every day (QD), and TAK-117 100 mg, capsule, orally, once on Monday, Wednesday and Friday each week (MWF QW) for up to 3 cycles (each cycle was 28 days), up to 10.4 weeks.
- Dose Escalation Treatment Arm A: Cohort 3A: TAK-228 2 mg, capsule (unmilled), orally, once daily every day (QD), and TAK-117 200 mg, capsule, orally, once on Monday, Wednesday and Friday each week (MWF QW) for up to 5 cycles (each cycle was 28 days), up to 21.0 weeks.
- Dose Escalation Treatment Arm A: Cohort 3A (Milled): TAK-228 2 mg, capsule (milled), orally, once daily every day (QD), and TAK-117 200 mg, capsule, orally, once on Monday, Wednesday and Friday each week (MWF QW) for up to 2 cycles (each cycle was 28 days), up to 6.1 weeks.
- Dose Escalation Treatment Arm A: Cohort 4A: TAK-228 2 mg, capsule (unmilled), orally, once daily every day (QD), and TAK-117 300 mg, capsule, orally, once on Monday, Wednesday and Friday each week (MWF QW) for up to 13 cycles (each cycle was 28 days), up to approximately 52 weeks.
- Dose Escalation Treatment Arm B: Cohort 1B: TAK-228 3 mg, capsule (unmilled), orally, once on Monday, Tuesday and Wednesday each week (MTuW QW), and TAK-117 100 mg, capsule, orally, once on MTuW QW for up to 6 cycles (each cycle was 28 days), up to 23.4 weeks.
- Dose Escalation Treatment Arm B: Cohort 2B: TAK-228 3 mg, capsule (unmilled), orally, once on Monday, Tuesday and Wednesday each week (MTuW QW), and TAK-117 200 mg, capsule, orally, once on MTuW QW for up to 6 cycles (each cycle was 28 days), up to 21.3 weeks.
- Dose Escalation Treatment Arm B: Cohort 3B: TAK-228 6 mg, capsule (unmilled), orally, once on Monday, Tuesday and Wednesday each week (MTuW QW), and TAK-117 200 mg, capsule, orally, once on MTuW QW for up to 5 cycles (each cycle was 28 days), up to 19.4 weeks.
- Dose Escalation Treatment Arm B: Cohort 3B (Milled): TAK-228 6 mg, capsule (milled), orally, once on Monday, Tuesday and Wednesday each week (MTuW QW), and TAK-117 200 mg, capsule, orally, once on MTuW QW for up to 4 cycles (each cycle was 28 days), up to 15.4 weeks.
- Dose Escalation Treatment Arm B: Cohort 4B: TAK-228 8 mg, capsule (unmilled), orally, once on Monday, Tuesday and Wednesday each week (MTuW QW), and TAK-117 200 mg, capsule, orally, once on MTuW QW for up to 2 cycles (each cycle was 28 days), up to 7.4 weeks.
- Dose Escalation Treatment Arm B: Cohort 5B (Milled): TAK-228 4 mg, capsule (milled), orally, once on Monday, Tuesday and Wednesday each week (MTuW QW), and TAK-117 200 mg, capsule, orally, once on MTuW QW for up to 9 cycles (each cycle was 28 days), up to 38.7 weeks.
- Dose Escalation Treatment Arm C: Cohort 1C: TAK-228 3 mg, capsule (unmilled), orally, once on MTuW QW, and TAK-117 400 mg, capsule, orally, once on MTuW QW for up to 17 cycles (each cycle was 28 days), up to 64.3 weeks.
- Dose Escalation Treatment Arm C: Cohort 2C (Milled): TAK-228 3 mg, capsule (milled), orally, once on MTuW QW, and TAK-117 300 mg, capsule, orally, once on MTuW QW for up to 11 cycles (each cycle was 28 days), up to 43.4 weeks.
- Drug-Drug Interaction (DDI) Expansion Cohort (Milled): TAK-228 4 mg, capsule (milled), orally, once on MTuW QW except on Days 15, 16 and 17 of Cycle 1, and TAK-117 200 mg, capsule, orally, once on MTuW QW except on Days 1, 2 and 3 of Cycle 1 for up to 8 cycles (each cycle was 28 days), up to approximately 31.4 weeks.
Period: Overall Study
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled) | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Started | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14 | 20
Completed (Completed=Participants who completed the study treatment.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14 | 20
Not completed — Progressive Disease | 4 | 0 | 3 | 0 | 3 | 1 | 1 | 1 | 4 | 3 | 12 | 5 | 8 | 17
Not completed — Adverse Event | 1 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 2 | 0 | 3 | 1 | 2 | 2
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Therapeutic Response | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all enrolled participants who received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled) | Drug-Drug Interaction (DDI) Expansion Cohort (Milled) | Total
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14 | 20 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (6.31) | 69.3 (5.13) | 50.6 (14.05) | 66.7 (5.86) | 48.7 (11.66) | 74.3 (5.13) | 69.3 (14.15) | 68.3 (9.24) | 58.0 (7.72) | 68.3 (4.16) | 56.6 (9.69) | 53.3 (14.36) | 56.5 (6.97) | 63.4 (9.10) | 59.4 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 7 | 3 | 2 | 1 | 2 | 1 | 4 | 2 | 11 | 2 | 7 | 13 | 64
  Male | 0 | 1 | 0 | 0 | 4 | 2 | 1 | 2 | 2 | 1 | 5 | 5 | 7 | 7 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 4 | 8
  Not Hispanic or Latino | 7 | 2 | 7 | 3 | 5 | 3 | 3 | 2 | 5 | 2 | 13 | 7 | 13 | 9 | 81
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 2 | 7 | 3 | 5 | 3 | 3 | 3 | 4 | 3 | 13 | 4 | 14 | 19 | 90
  Black Or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 5
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 1 | 2 | 1 | 11
  Spain | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 3 | 1 | 5 | 1 | 4 | 12 | 31
  United States | 7 | 3 | 6 | 3 | 3 | 3 | 2 | 1 | 2 | 1 | 8 | 5 | 8 | 7 | 59
Height [Mean (Standard Deviation); unit: cm] | 164.0 (3.84) | 165.1 (5.08) | 161.6 (3.26) | 159.4 (7.73) | 169.8 (8.73) | 169.0 (12.86) | 157.3 (4.25) | 168.5 (15.02) | 168.3 (12.41) | 168.5 (8.30) | 168.7 (11.24) | 180.7 (9.35) | 170.7 (7.86) | 163.7 (7.64) | 167.3 (9.67)
Weight [Mean (Standard Deviation); unit: kg] | 63.8 (9.11) | 78.4 (1.34) | 69.7 (14.20) | 49.8 (8.06) | 79.5 (19.91) | 67.6 (20.33) | 62.5 (15.32) | 73.7 (17.32) | 78.2 (22.65) | 79.3 (9.11) | 71.4 (13.00) | 79.9 (15.19) | 78.6 (17.55) | 64.6 (12.08) | 71.4 (15.63)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated as weight/[height^2].
  kg/m^2 | 23.7 (2.80) | 28.8 (2.09) | 26.7 (5.65) | 19.9 (5.06) | 27.3 (5.09) | 23.2 (3.36) | 25.4 (7.18) | 26.2 (6.76) | 27.2 (4.60) | 27.9 (3.11) | 25.2 (4.30) | 24.3 (3.27) | 27.0 (5.74) | 24.1 (4.06) | 25.4 (4.66)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One or More Treatment-Emergent Adverse Event (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. A SAE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above-mentioned criteria.
Time Frame: From Baseline to 30 days after the last dose of study drug (Up to approximately 68 weeks)
Population: Safety population consisted of all enrolled participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled) | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14 | 20
Participants
  AEs | 7 | 3 | 7 | 3 | 5 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14 | 19
  SAEs | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 4 | 4 | 6 | 9

2. Primary Outcome: Tmax: Time to Reach the Maximum Observed Plasma Concentration After Single-dose and Multiple-dose of TAK-228 in the Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: Pharmacokinetic (PK) population consisted of all participants enrolled in the study who received at least 1 dose of TAK-228 and TAK-117 and had sufficient concentration-time data to calculate 1 or more PK parameters. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Median (Full Range); unit: hour
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
hour
  Cycle 1, Day 1: number analyzed (Participants) | 7 | 3 | 7 | 3 | 5 | 3 | 3 | 3 | 6 | 3 | 16 | 6 | 14
  Cycle 1, Day 1 | 1.000 [0.50 to 4.00] | 1.000 [0.97 to 1.03] | 1.000 [0.50 to 4.07] | 2.050 [0.53 to 2.07] | 1.033 [1.00 to 2.08] | 2.083 [1.97 to 4.02] | 1.000 [0.48 to 1.07] | 1.067 [1.03 to 8.12] | 1.358 [0.50 to 4.00] | 1.067 [0.98 to 3.83] | 1.000 [0.50 to 2.15] | 0.725 [0.43 to 2.08] | 0.983 [0.47 to 4.17]
  Cycle 1, Day 24: number analyzed (Participants) | 6 | 2 | 6 | 0 | 5 | 3 | 2 | 3 | 4 | 1 | 9 | 4 | 11
  Cycle 1, Day 24 | 1.000 [0.50 to 2.00] | 0.758 [0.48 to 1.03] | 1.400 [0.45 to 4.08] |  | 2.000 [0.92 to 2.25] | 4.000 [1.00 to 4.12] | 1.408 [1.00 to 1.82] | 0.617 [0.48 to 2.00] | 0.925 [0.50 to 2.15] | 4.000 [4.000 to 4.000] | 1.033 [0.47 to 2.30] | 2.083 [1.95 to 4.87] | 1.017 [0.50 to 7.03]

3. Primary Outcome: Cmax: Maximum Observed Plasma Concentration After Single-dose and Multiple-dose of TAK-228 in the Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: PK population consisted of all participants enrolled in the study who received at least 1 dose of TAK-228 and TAK-117 and had sufficient concentration-time data to calculate 1 or more PK parameters. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 7 | 3 | 7 | 3 | 5 | 3 | 3 | 3 | 6 | 3 | 16 | 6 | 14
  Cycle 1, Day 1 | 24.63 (7.355) | 39.73 (7.853) | 25.80 (8.188) | 28.67 (3.702) | 18.26 (8.610) | 21.69 (29.273) | 48.90 (28.157) | 33.30 (16.301) | 53.10 (7.257) | 53.53 (29.788) | 42.17 (11.495) | 27.53 (11.665) | 26.51 (12.788)
  Cycle 1, Day 24: number analyzed (Participants) | 6 | 2 | 6 | 0 | 5 | 3 | 2 | 3 | 4 | 1 | 9 | 4 | 11
  Cycle 1, Day 24 | 27.78 (6.632) | 53.55 (2.192) | 29.45 (9.746) |  | 13.75 (6.938) | 37.36 (49.078) | 46.10 (17.253) | 72.43 (13.094) | 61.58 (14.894) | 17.1 (0) | 50.68 (12.055) | 17.75 (4.865) | 35.59 (18.415)

4. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Observed Quantifiable Concentration After Single-dose and Multiple-dose of TAK-228 in the Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
ng*hr/mL
  Cycle 1, Day 1: number analyzed (Participants) | 7 | 3 | 7 | 3 | 5 | 3 | 3 | 3 | 6 | 3 | 16 | 6 | 14
  Cycle 1, Day 1 | 120.888 (36.1184) | 247.361 (156.0211) | 138.929 (37.3727) | 230.983 (14.6292) | 109.622 (45.6613) | 126.062 (120.8204) | 303.897 (152.5659) | 287.283 (268.7088) | 351.602 (122.6407) | 382.588 (250.2623) | 249.341 (128.4868) | 168.408 (103.9245) | 160.670 (90.6815)
  Cycle 1, Day 24: number analyzed (Participants) | 6 | 2 | 6 | 0 | 5 | 3 | 2 | 3 | 4 | 1 | 9 | 4 | 11
  Cycle 1, Day 24 | 206.418 (169.5373) | 208.389 (78.6461) | 200.762 (56.1368) |  | 115.884 (50.7913) | 203.836 (120.1336) | 410.604 (265.8768) | 535.365 (256.8762) | 331.286 (133.7879) | 305.97 (0) | 317.111 (151.6045) | 132.058 (71.7154) | 211.792 (100.9091)

5. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) After Single-dose and Multiple-dose of TAK-228 in the Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
hour
  Cycle 1, Day 1: number analyzed (Participants) | 5 | 3 | 5 | 3 | 4 | 1 | 3 | 1 | 4 | 2 | 14 | 6 | 5
  Cycle 1, Day 1 | 5.090 (2.1653) | 5.783 (3.3941) | 6.214 (2.6649) | 7.450 (0.7368) | 6.975 (1.0108) | 4.65 (0) | 8.412 (1.3996) | 4.96 (0) | 5.792 (3.4405) | 6.799 (5.5740) | 6.320 (1.7839) | 5.512 (2.1598) | 7.593 (1.1365)
  Cycle 1, Day 24: number analyzed (Participants) | 5 | 2 | 5 | 0 | 3 | 1 | 1 | 3 | 3 | 0 | 8 | 1 | 9
  Cycle 1, Day 24 | 5.489 (2.4782) | 4.686 (2.1265) | 5.521 (1.6417) |  | 7.635 (1.1253) | 5.43 (0) | 8.5 (0) | 6.808 (1.7326) | 6.221 (1.0591) |  | 5.940 (1.6737) | 6.42 (0) | 6.354 (1.9320)

6. Primary Outcome: CL/F: Apparent Clearance After Extravascular Administration, Calculated Using the Observed Value of the Last Quantifiable Concentration After Single-dose and Multiple-dose of TAK-228 in the Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: PK population consisted of all participants enrolled during the dose escalation and expansion stage of the study who received at least 1 dose of TAK-228 and TAK-117 and had sufficient concentration-time data to calculate 1 or more PK parameters. Number analyzed is the number of participants who were evaluable at each category.
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
L/hour
  Cycle 1, Day 1: number analyzed (Participants) | 5 | 3 | 5 | 3 | 4 | 1 | 3 | 1 | 4 | 2 | 14 | 6 | 5
  Cycle 1, Day 1 | 16.534 (5.4762) | 19.049 (11.8558) | 14.419 (7.5636) | 7.694 (0.5750) | 15.311 (3.6762) | 11.38 (0) | 10.728 (6.9669) | 28.54 (0) | 19.999 (10.0509) | 16.259 (9.3725) | 17.924 (9.5261) | 22.715 (14.7252) | 13.933 (5.4880)
  Cycle 1, Day 24: number analyzed (Participants) | 5 | 2 | 5 | 0 | 6 | 1 | 1 | 3 | 3 | 0 | 8 | 1 | 9
  Cycle 1, Day 24 | 14.720 (4.5824) | 18.207 (4.1819) | 10.597 (3.9917) |  | 15.683 (2.9149) | 9.23 (0) | 13.58 (0) | 12.817 (4.7929) | 19.060 (7.1913) |  | 14.196 (5.3137) | 15.53 (0) | 16.133 (8.6701)

7. Primary Outcome: RAC: Accumulation Ratio for TAK-228 in the Dose Escalation Cohort
Description: Accumulation ratio was based on AUC(0-24) between Cycle 1 Day 24 and Cycle 1 Day 1 (e.g. AUC(0-24) [Cycle 1 Day 24]/ AUC(0-24) [Cycle1 Day 1].
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: PK population consisted of all participants enrolled in the study who received at least 1 dose of TAK-228 and TAK-117 and had sufficient concentration-time data to calculate 1 or more PK parameters. Overall number of participants analyzed is the number of participants with evaluable data at both Days 1 and 24.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 3 | 1 | 4 | 0 | 3 | 2 | 2 | 2 | 2 | 1 | 8 | 2 | 6
ratio | 2.225 (1.4576) | 1.25 (0) | 1.495 (0.1884) |  | 1.219 (0.3497) | 1.569 (0.4099) | 1.712 (0.2650) | 1.718 (0.4329) | 1.015 (0.1453) | 1.58 (0) | 1.172 (0.3363) | 1.213 (0.1306) | 1.461 (0.2246)

8. Primary Outcome: Peak to Trough Ratio for TAK-228 After Single-dose and Multiple-dose of TAK-228 in the Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
ratio
  Cycle 1, Day 1: number analyzed (Participants) | 4 | 2 | 5 | 3 | 4 | 2 | 3 | 2 | 5 | 2 | 14 | 4 | 9
  Cycle 1, Day 1 | 16.546 (6.5659) | 13.588 (8.3649) | 14.553 (6.8807) | 10.420 (1.5662) | 13.983 (6.6782) | 23.757 (31.1525) | 14.336 (7.0986) | 20.212 (22.0357) | 13.227 (8.3834) | 5.761 (1.5250) | 22.676 (14.2142) | 15.012 (6.5253) | 10.725 (2.7876)
  Cycle 1, Day 24: number analyzed (Participants) | 4 | 1 | 5 | 0 | 4 | 3 | 2 | 3 | 6 | 1 | 8 | 2 | 9
  Cycle 1, Day 24 | 12.145 (6.0465) | 27.66 (0) | 14.691 (8.1076) |  | 9.363 (6.6336) | 21.864 (33.1541) | 9.305 (4.7969) | 21.979 (13.7911) | 31.971 (19.6410) | 1.8 (0) | 22.555 (10.4006) | 8.805 (7.3805) | 21.157 (14.9668)

9. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) After Single-dose and Multiple-dose of TAK-117 in the Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
hour
  Cycle 1, Day 1: number analyzed (Participants) | 6 | 3 | 7 | 3 | 6 | 1 | 3 | 3 | 6 | 3 | 16 | 7 | 14
  Cycle 1, Day 1 | 0.800 [0.50 to 2.03] | 2.000 [1.03 to 2.00] | 2.050 [0.52 to 4.08] | 2.050 [1.03 to 2.07] | 3.017 [1.85 to 7.50] | 1.97 [1.97 to 1.97] | 2.000 [1.07 to 4.18] | 1.033 [0.50 to 8.12] | 4.008 [0.50 to 7.25] | 3.883 [2.42 to 7.33] | 1.925 [1.00 to 4.15] | 2.083 [0.95 to 6.03] | 3.125 [0.50 to 22.58]
  Cycle 1, Day 24: number analyzed (Participants) | 6 | 2 | 6 | 0 | 5 | 3 | 3 | 3 | 4 | 1 | 9 | 4 | 11
  Cycle 1, Day 24 | 1.000 [0.55 to 4.00] | 1.025 [1.02 to 1.03] | 4.108 [0.93 to 8.02] |  | 2.417 [1.97 to 4.00] | 2.000 [1.92 to 4.00] | 1.408 [1.00 to 1.82] | 0.883 [0.62 to 4.05] | 3.150 [2.00 to 7.02] | 7.33 [7.33 to 7.33] | 2.000 [1.00 to 8.02] | 2.050 [1.40 to 4.27] | 1.117 [0.95 to 8.07]

10. Primary Outcome: Cmax: Maximum Observed Plasma Concentration After Single-dose and Multiple-dose of TAK-117 in the Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 6 | 3 | 7 | 3 | 6 | 1 | 3 | 3 | 6 | 3 | 16 | 7 | 14
  Cycle 1, Day 1 | 1800.0 (1049.25) | 988.7 (858.57) | 3067.1 (1243.50) | 4950.0 (3381.06) | 4136.7 (1487.68) | 2420 (0) | 3836.7 (656.07) | 1631.3 (1305.25) | 2711.7 (1172.97) | 2568.7 (2107.04) | 3369.4 (1417.31) | 3077.7 (1629.05) | 3353.0 (1955.02)
  Cycle 1, Day 24: number analyzed (Participants) | 6 | 2 | 6 | 0 | 5 | 3 | 2 | 3 | 4 | 1 | 9 | 4 | 11
  Cycle 1, Day 24 | 2514.0 (1597.13) | 2720.0 (1286.93) | 3438.3 (1687.00) |  | 3624.0 (2925.79) | 1054.8 (1454.94) | 6180.0 (127.28) | 4876.7 (848.84) | 4477.5 (953.88) | 100 (0) | 4863.3 (1142.54) | 3755.0 (2831.78) | 4805.3 (2893.99)

11. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Observed Quantifiable Concentration After Single-dose and Multiple-dose of TAK-117 in Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
ng*hr/mL
  Cycle 1, Day 1: number analyzed (Participants) | 6 | 3 | 7 | 3 | 6 | 1 | 3 | 3 | 6 | 3 | 16 | 7 | 14
  Cycle 1, Day 1 | 14586.139 (10434.5445) | 11550.908 (11672.0852) | 43948.190 (25421.3428) | 69617.994 (46233.0898) | 54993.211 (27446.4517) | 26746.78 (0) | 47803.262 (4758.7418) | 23148.610 (27836.8878) | 38563.109 (23484.8077) | 39903.517 (33243.1212) | 38224.835 (22368.0163) | 30925.255 (15126.4913) | 46451.606 (33137.8861)
  Cycle 1, Day 24: number analyzed (Participants) | 6 | 2 | 6 | 0 | 5 | 3 | 2 | 3 | 4 | 1 | 9 | 4 | 11
  Cycle 1, Day 24 | 31723.844 (38363.4872) | 22566.251 (13562.8900) | 50960.181 (32295.5320) |  | 46278.615 (48171.7982) | 12428.783 (16745.7861) | 90462.795 (14090.4676) | 67186.097 (49493.0584) | 55908.919 (39888.9699) | 1674.23 (0) | 72432.560 (27615.6802) | 46164.679 (37938.0208) | 70490.572 (58515.7794)

12. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) After Single-dose and Multiple-dose of TAK-117 in Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
hour
  Cycle 1, Day 1: number analyzed (Participants) | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 4 | 3 | 2
  Cycle 1, Day 1 | 6.590 (3.4673) | 4.92 (0) |  |  |  |  |  | 3.839 (3.5498) | 7.465 (2.2023) |  | 4.858 (2.7928) | 6.379 (1.5369) | 7.368 (0.3774)
  Cycle 1, Day 24: number analyzed (Participants) | 4 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 3 | 2 | 5
  Cycle 1, Day 24 | 5.722 (3.1259) | 6.53 (0) | 2.98 (0) |  | 3.2 (0) | 8.37 (0) |  | 6.233 (4.4813) | 4.61 (0) |  | 7.717 (2.6428) | 5.853 (2.1534) | 5.984 (3.6558)

13. Primary Outcome: CL/F: Apparent Clearance After Extravascular Administration, Calculated Using the Observed Value of the Last Quantifiable Concentration After Single-dose and Multiple-dose of TAK-117 in Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
L/hr
  Cycle 1, Day 1: number analyzed (Participants) | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 4 | 3 | 2
  Cycle 1, Day 1 | 16.993 (23.6496) | 9.79 (0) |  |  |  |  |  | 194.998 (258.2751) | 20.944 (16.6625) |  | 17.879 (17.8072) | 21.075 (16.4116) | 32.455 (35.8687)
  Cycle 1, Day 24: number analyzed (Participants) | 4 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 3 | 2 | 5
  Cycle 1, Day 24 | 13.821 (16.5047) | 7.18 (0) | 17.95 (0) |  | 9.25 (0) | 19.7 (0) |  | 5.328 (1.2794) | 5.45 (0) |  | 4.803 (2.7599) | 11.199 (8.4334) | 67.750 (110.0873)

14. Primary Outcome: RAC: Accumulation Ratio for TAK-117 in the Dose Escalation Cohort
Description: as for outcome 7
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 4 | 1 | 5 | 0 | 5 | 1 | 2 | 2 | 3 | 1 | 9 | 3 | 9
ratio | 0.965 (0.1423) | 1.33 (0) | 1.161 (0.2506) |  | 1.049 (0.9033) | 1.18 (0) | 2.007 (0.4766) | 2.687 (0.5700) | 1.748 (1.1575) | 0.91 (0) | 1.879 (1.5772) | 0.925 (0.6281) | 4.183 (5.8060)

15. Primary Outcome: Peak to Trough Ratio After Single-dose and Multiple-dose of TAK-117 in Dose Escalation Cohort
Time Frame: Cycle 1: Days 1 and 24 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14
ratio
  Cycle 1, Day 1: number analyzed (Participants) | 5 | 2 | 6 | 3 | 6 | 1 | 3 | 2 | 6 | 3 | 13 | 6 | 13
  Cycle 1, Day 1 | 20.138 (21.6013) | 8.845 (7.8516) | 2.551 (0.9673) | 2.676 (0.1635) | 4.373 (3.3285) | 3.93 (0) | 3.602 (0.8361) | 6.640 (7.3746) | 6.877 (8.8600) | 2.631 (0.5993) | 6.872 (8.3680) | 11.494 (10.9430) | 3.426 (2.3804)
  Cycle 1, Day 24: number analyzed (Participants) | 5 | 2 | 5 | 0 | 5 | 3 | 2 | 3 | 3 | 1 | 9 | 4 | 9
  Cycle 1, Day 24 | 10.023 (9.0435) | 11.256 (7.1426) | 2.294 (0.5975) |  | 20.124 (33.8991) | 3.931 (2.4369) | 3.464 (0.1399) | 54.242 (87.1445) | 11.832 (15.4766) | 1.96 (0) | 5.482 (6.7075) | 11.184 (8.0869) | 4.664 (3.9973)

16. Primary Outcome: Tmax: Time to Reach the Maximum Observed Plasma Concentration for TAK-228 in DDI Expansion Cohort
Time Frame: Cycle 1, Day 3 predose and at multiple timepoints (up to 8 hours) postdose; Cycle 1, Day 10 predose and at multiple timepoints (up to 24 hours) postdose
Population: PK DDI-evaluable population consisted of all participants from Expansion Phase with sufficient dosing and concentration-time PK data to reliably estimate PK parameters for statistical analyses of effect of TAK-228 on TAK-117 PK and effect of TAK-117 on TAK-228 PK. Number analyzed is number of participants with evaluable data at given time-point.
Measure: Median (Full Range); unit: hour
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
hour
  Cycle 1, Day 3, TAK-228 administered alone: number analyzed (Participants) | 19
  Cycle 1, Day 3, TAK-228 administered alone | 1.000 [0.38 to 4.08]
  Cycle 1, Day 10, TAK-228 administered with TAK-117: number analyzed (Participants) | 19
  Cycle 1, Day 10, TAK-228 administered with TAK-117 | 0.983 [0.42 to 2.02]

17. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-228 in DDI Expansion Cohort
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
ng/mL
  Cycle 1, Day 3, TAK-228 administered alone: number analyzed (Participants) | 19
  Cycle 1, Day 3, TAK-228 administered alone | 60.02 (21.808)
  Cycle 1, Day 10, TAK-228 administered with TAK-117: number analyzed (Participants) | 19
  Cycle 1, Day 10, TAK-228 administered with TAK-117 | 71.99 (22.546)

18. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Observed Quantifiable Concentration for TAK-228 in DDI Expansion Cohort
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
ng*hr/mL
  Cycle 1, Day 3, TAK-228 administered alone: number analyzed (Participants) | 19
  Cycle 1, Day 3, TAK-228 administered alone | 301.613 (123.9584)
  Cycle 1, Day 10, TAK-228 administered with TAK-117: number analyzed (Participants) | 19
  Cycle 1, Day 10, TAK-228 administered with TAK-117 | 390.307 (155.3378)

19. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) for TAK-228 in DDI Expansion Cohort
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
hour
  Cycle 1, Day 3, TAK-228 administered alone: number analyzed (Participants) | 15
  Cycle 1, Day 3, TAK-228 administered alone | 6.823 (2.1608)
  Cycle 1, Day 10, TAK-228 administered with TAK-117: number analyzed (Participants) | 16
  Cycle 1, Day 10, TAK-228 administered with TAK-117 | 6.546 (1.8351)

20. Primary Outcome: CL/F: Apparent Clearance After Extravascular Administration, Calculated Using the Observed Value of the Last Quantifiable Concentration for TAK-228 in DDI Expansion Cohort
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: L/hour
Groups:
- Drug-Drug Interaction (DDI) Expansion Cohort (Milled)): TAK-228 4 mg, capsule (milled), orally, once on MTuW QW except on Days 15, 16 and 17 of Cycle 1, and TAK-117 200 mg, capsule, orally, once on MTuW QW except on Days 1, 2 and 3 of Cycle 1 for up to 8 cycles (each cycle was 28 days), up to approximately 31.4 weeks.
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled))
Number analyzed (Participants) | 20
L/hour
  Cycle 1, Day 3, TAK-228 administered alone: number analyzed (Participants) | 15
  Cycle 1, Day 3, TAK-228 administered alone | 15.368 (10.9714)
  Cycle 1, Day 10, TAK-228 administered with TAK-117: number analyzed (Participants) | 16
  Cycle 1, Day 10, TAK-228 administered with TAK-117 | 13.359 (11.3718)

21. Primary Outcome: Peak to Trough Ratio for TAK-228 in DDI Expansion Cohort
Time Frame: as for outcome 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
ratio
  Cycle 1, Day 3, TAK-228 administered alone: number analyzed (Participants) | 17
  Cycle 1, Day 3, TAK-228 administered alone | 22.982 (11.6286)
  Cycle 1, Day 10, TAK-228 administered with TAK-117: number analyzed (Participants) | 18
  Cycle 1, Day 10, TAK-228 administered with TAK-117 | 23.931 (15.6395)

22. Primary Outcome: Tmax: Time to Reach the Maximum Observed Plasma Concentration for TAK-117 in DDI Expansion Cohort
Time Frame: Cycle 1, Day 3 predose and at multiple timepoints (up to 8 hours) postdose; Cycle 1, Day 17 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 16
Measure: Median (Full Range); unit: hour
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
hour
  Cycle 1, Day 10, TAK-117 administered with TAK-228: number analyzed (Participants) | 19
  Cycle 1, Day 10, TAK-117 administered with TAK-228 | 1.033 [0.50 to 4.12]
  Cycle 1, Day 17, TAK-117 administered alone: number analyzed (Participants) | 19
  Cycle 1, Day 17, TAK-117 administered alone | 1.983 [0.50 to 7.25]

23. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-117 in DDI Expansion Cohort
Time Frame: as for outcome 22
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
ng/mL
  Cycle 1, Day 10, TAK-117 administered with TAK-228: number analyzed (Participants) | 19
  Cycle 1, Day 10, TAK-117 administered with TAK-228 | 5357.3 (2842.40)
  Cycle 1, Day 17, TAK-117 administered alone: number analyzed (Participants) | 19
  Cycle 1, Day 17, TAK-117 administered alone | 5332.6 (2955.51)

24. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Observed Quantifiable Concentration for TAK-117 in DDI Expansion Cohort
Time Frame: as for outcome 22
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
ng*hr/mL
  Cycle 1, Day 10, TAK-117 administered with TAK-228: number analyzed (Participants) | 19
  Cycle 1, Day 10, TAK-117 administered with TAK-228 | 61148.949 (42799.7918)
  Cycle 1, Day 17, TAK-117 administered alone: number analyzed (Participants) | 19
  Cycle 1, Day 17, TAK-117 administered alone | 63975.156 (53764.5716)

25. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) for TAK-117 in DDI Expansion Cohort
Time Frame: as for outcome 22
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
hour
  Cycle 1, Day 10, TAK-117 administered with TAK-228: number analyzed (Participants) | 8
  Cycle 1, Day 10, TAK-117 administered with TAK-228 | 6.420 (2.3635)
  Cycle 1, Day 17, TAK-117 administered alone: number analyzed (Participants) | 11
  Cycle 1, Day 17, TAK-117 administered alone | 5.717 (2.3715)

26. Primary Outcome: CL/F: Apparent Clearance After Extravascular Administration, Calculated Using the Observed Value of the Last Quantifiable Concentration for TAK-117 in DDI Expansion Cohort
Time Frame: as for outcome 22
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
L/hour
  Cycle 1, Day 10, TAK-117 administered with TAK-228: number analyzed (Participants) | 8
  Cycle 1, Day 10, TAK-117 administered with TAK-228 | 11.797 (18.0040)
  Cycle 1, Day 17, TAK-117 administered alone: number analyzed (Participants) | 11
  Cycle 1, Day 17, TAK-117 administered alone | 9.134 (8.7741)

27. Primary Outcome: Peak to Trough Ratio for TAK-117 in DDI Expansion Cohort
Time Frame: as for outcome 22
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 20
ratio
  Cycle 1, Day 10, TAK-117 administered with TAK-228: number analyzed (Participants) | 17
  Cycle 1, Day 10, TAK-117 administered with TAK-228 | 7.423 (7.423)
  Cycle 1, Day 17, TAK-117 administered alone: number analyzed (Participants) | 18
  Cycle 1, Day 17, TAK-117 administered alone | 21.357 (44.3461)

28. Secondary Outcome: Objective Response Rate (ORR) Based on Investigator's Assessment According to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR defined as the percentage of participants with Complete Response (CR) + Partial Response (PR) as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 for target lesions and assessed by CT or MRI. CR is defined as disappearance of all target lesions and PR is defined as 30% decrease in the sum of the longest diameter (LD) of target lesions. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline, Days 22 up to Day 28 of Cycle and every even-numbered cycle until disease progression or EOS (Up to approximately 68 weeks)
Population: Safety population consisted of all enrolled participants who received at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled) | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 7 | 3 | 7 | 3 | 6 | 3 | 3 | 3 | 6 | 3 | 16 | 7 | 14 | 20
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 20.0

29. Secondary Outcome: Duration of Response (DOR)
Description: The DOR is defined as the time from the date of first documented response of CR/PR to the first documented progressive disease (PD), or censored at the last response assessment date that is SD or better for a participant that has not progressed. CR was defined as the disappearance of all target lesions and for non-target lesions, the disappearance of all non-target lesions and normalization of tumor marker level. PR was defined of at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD and for non-target lesions.
Time Frame: as for outcome 28
Population: Safety population consisted of all enrolled participants who received at least 1 dose of any study drug. Data for this outcome measure is reported for the participants with objective response available.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled) | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
days |  |  |  |  |  |  |  |  |  |  |  |  |  | 92 [1 to 288]

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose of study drug (Up to approximately 68 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dose Escalation Treatment Arm A: Cohort 1A | Dose Escalation Treatment Arm A: Cohort 2A | Dose Escalation Treatment Arm A: Cohort 3A | Dose Escalation Treatment Arm A: Cohort 3A (Milled) | Dose Escalation Treatment Arm A: Cohort 4A | Dose Escalation Treatment Arm B: Cohort 1B | Dose Escalation Treatment Arm B: Cohort 2B | Dose Escalation Treatment Arm B: Cohort 3B | Dose Escalation Treatment Arm B: Cohort 3B (Milled) | Dose Escalation Treatment Arm B: Cohort 4B | Dose Escalation Treatment Arm B: Cohort 5B (Milled) | Dose Escalation Treatment Arm C: Cohort 1C | Dose Escalation Treatment Arm C: Cohort 2C (Milled) | Drug-Drug Interaction (DDI) Expansion Cohort (Milled)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3 | 1/7 | 0/3 | 1/6 | 0/3 | 0/3 | 0/3 | 0/6 | 0/3 | 2/16 | 0/7 | 0/14 | 2/20
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/3 | 1/7 | 1/3 | 1/6 | 0/3 | 1/3 | 1/3 | 1/6 | 1/3 | 4/16 | 4/7 | 6/14 | 9/20
Other Adverse Events (participants affected / at risk) | 6/7 | 3/3 | 7/7 | 3/3 | 5/6 | 3/3 | 3/3 | 3/3 | 6/6 | 3/3 | 16/16 | 7/7 | 13/14 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Treatment Arm A: Cohort 1A (N=7) | Dose Escalation Treatment Arm A: Cohort 2A (N=3) | Dose Escalation Treatment Arm A: Cohort 3A (N=7) | Dose Escalation Treatment Arm A: Cohort 3A (Milled) (N=3) | Dose Escalation Treatment Arm A: Cohort 4A (N=6) | Dose Escalation Treatment Arm B: Cohort 1B (N=3) | Dose Escalation Treatment Arm B: Cohort 2B (N=3) | Dose Escalation Treatment Arm B: Cohort 3B (N=3) | Dose Escalation Treatment Arm B: Cohort 3B (Milled) (N=6) | Dose Escalation Treatment Arm B: Cohort 4B (N=3) | Dose Escalation Treatment Arm B: Cohort 5B (Milled) (N=16) | Dose Escalation Treatment Arm C: Cohort 1C (N=7) | Dose Escalation Treatment Arm C: Cohort 2C (Milled) (N=14) | Drug-Drug Interaction (DDI) Expansion Cohort (Milled) (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with DDI expansion cohort (milled) and is not related.
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with dose escalation treatment arm A: cohort 4A and is not related.
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with dose escalation treatment arm A: cohort 5B (milled) and is not related.
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with DDI expansion cohort (milled) and is not related.
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with dose escalation treatment arm A: cohort 5B (milled) and is not related.
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with dose escalation treatment arm A: cohort 3A and is not related.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Treatment Arm A: Cohort 1A (N=7) | Dose Escalation Treatment Arm A: Cohort 2A (N=3) | Dose Escalation Treatment Arm A: Cohort 3A (N=7) | Dose Escalation Treatment Arm A: Cohort 3A (Milled) (N=3) | Dose Escalation Treatment Arm A: Cohort 4A (N=6) | Dose Escalation Treatment Arm B: Cohort 1B (N=3) | Dose Escalation Treatment Arm B: Cohort 2B (N=3) | Dose Escalation Treatment Arm B: Cohort 3B (N=3) | Dose Escalation Treatment Arm B: Cohort 3B (Milled) (N=6) | Dose Escalation Treatment Arm B: Cohort 4B (N=3) | Dose Escalation Treatment Arm B: Cohort 5B (Milled) (N=16) | Dose Escalation Treatment Arm C: Cohort 1C (N=7) | Dose Escalation Treatment Arm C: Cohort 2C (Milled) (N=14) | Drug-Drug Interaction (DDI) Expansion Cohort (Milled) (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 2 | 6 | 3 | 4 | 1 | 3 | 3 | 5 | 3 | 11 | 4 | 10 | 11
Vomiting (Gastrointestinal disorders) | 1 | 1 | 5 | 2 | 3 | 0 | 2 | 2 | 4 | 3 | 8 | 2 | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 3 | 1 | 2 | 2 | 2 | 1 | 2 | 2 | 6 | 3 | 7 | 6
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 7
Constipation (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 3 | 3 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2
Oral pain (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 3 | 1 | 3 | 3 | 2 | 1 | 2 | 2 | 6 | 2 | 6 | 4
Asthenia (General disorders) | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 4 | 10
Oedema peripheral (General disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 1 | 3 | 2
Chills (General disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 3 | 1 | 3 | 2 | 0 | 1 | 3 | 1 | 1 | 1 | 3 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2 | 1 | 3 | 2 | 0 | 1 | 3 | 1 | 1 | 1 | 2 | 2
Weight decreased (Investigations) | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 2
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 2 | 2 | 2 | 1 | 2 | 2 | 1 | 2 | 2 | 0 | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 4 | 1 | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 2 | 0 | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 3 | 3 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 3
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness Transitory (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear Discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Dry Eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye Oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal Incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorectal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tongue Oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gait Disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Early Satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hernia Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion Site Extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Medical Device Site Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture Site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temperature Intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Unevaluable Event (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture Site Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Disorder Postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stoma Site Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram Qt Prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Albumin Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Cholesterol Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Sodium Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Restless Legs Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Speech Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vocal Cord Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Libido Decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary Hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Breast Oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast Tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal Burning Sensation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vena Cava Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Venous Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acne Cystic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT01899053/SAP_000.pdf
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT01899053/Prot_001.pdf